CLINICAL TRIAL: NCT02171572
Title: Safety, Tolerability and Pharmacokinetics Study After Single and Multiple Oral Doses of Dabigatran Etexilate Capsule (110mg,150 mg b.i.d., 7 Days) in Healthy Chinese Subjects (Open Label Study)
Brief Title: Single and Multiple Oral Doses of Dabigatran Etexilate in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.81
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- Dabigatran etexilate low (Experimental)
  Interventions: Drug: Dabigatran etexilate low
- Dabigatran etexilate high (Experimental)
  Interventions: Drug: Dabigatran etexilate high

INTERVENTIONS:
Drug: Dabigatran etexilate low
  Arms: Dabigatran etexilate low
Drug: Dabigatran etexilate high
  Arms: Dabigatran etexilate high

SUMMARY:
The objective of the current study is to investigate safety, tolerability and, pharmacokinetics of dabigatran etexilate following oral administration of single and multiple oral doses (110mg, 150 mg b.i.d., 7 days) in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR and body temperature), 12-lead ECG, clinical laboratory tests

  * No finding of clinical relevance.
  * No evidence of a clinically relevant concomitant disease.
* Age: ≥18 and ≤45 years.
* Body Mass Index (BMI): ≥18 and <25 kg/m2.
* Signed and dated written informed consent prior to admission to the trial in accordance with Chinese GCP.

Exclusion Criteria:

* Current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Subject can not use an adequate form of contraception from the time of the first dose on Day 1 up to end-of study examination.
* Current diseases of the central nervous system (such as epilepsy), or psychiatric disorders or neurological disorders.
* History of clinically significant orthostatic hypotension, clinically significant current or past fainting spells or blackouts.
* Chronic or relevant acute infections.
* History of

  * allergy/hypersensitivity (including drug allergy) which was deemed relevant to the safety assessment as judged by the investigator (excluding asymptomatic seasonal rhinitis/hay fever)
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic diseases.
  * cerebral bleeding (e.g. after a car accident).
  * concussions (head trauma resulting in injuring to brain) with or without loss of consciousness.
* Intake of drugs with a long half-life (> 24 hours) within at least 1 month or less than 10 half-lives, whichever was shorter, of the respective drug prior to administration or during the trial.
* Use of aspirin (including over-the-counter medications), antiplatelet agents like ticlopidine or dipyridamole, chronic administration of non-steroidal anti-inflammatory drugs (NSAID), coumadin like anticoagulants, chronic use of corticosteroids, heparin or fibrinolytic agents within 14 days prior to administration up to end-of-study examination.
* Participation in another trial with an investigational drug within 3 months prior to administration up to end-of-study examination.
* Smoker (>10 cigarettes/day or inability to refrain from smoking during the trial).
* Alcohol abuse (more than 60 g/day; confirmed by interview).
* Drug abuse (confirmed by interview).
* Blood donation (more than 100 mL from 3 months prior to screening and any blood donation from screening up to end-of-study examination).
* Excessive physical activities (within 7 days prior to the first drug administration up to end-of-study examination).
* Any laboratory value outside the reference range that is of clinical relevance.
* Known hypersensitivity to the investigational drug or its excipients.
* Subject who was judged ineligible by the investigator or the sub-investigator.
* History of any familial bleeding disorder.
* Thrombocytes < 100×109 .
* Pregnant female subjects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Changes in physical examination | Day 1 and 14
Changes in vital signs | Day 1 to 14
Changes in 12-lead electrocardiogram (ECG) | Day 1, Day 4-10, day 14
Changes from baseline in laboratory examinations | Day 1, 2, 4, 7, 11, 14
Occurrence of adverse events | up to 7 days after last drug intake

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the single dose on Day 1) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
AUC 0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
AUC0-∞ (amount of analyte that is eliminated in area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
λz (terminal rate constant in plasma) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
t1/2, (terminal half-life of the analyte in plasma) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
MRTpo, (mean residence time of the analyte in the body after oral administration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
CL/F, (apparent clearance of the analyte in plasma following extravascular administration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular administration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after single dose of study drug
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
λz,ss (terminal rate constant in plasma at steady state) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
CL/F,ss (apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
RA,Cmax, (calculated as Cmax,ss/Cmax) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
RA,AUC, (calculated as AUCτ,ss/AUCτ,1) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug
linearity index (LI) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours after last multiple dose of study drug